# **Study Protocol**

Alcohol Health Education With Personalized Feedback Boosters

NCT03440463

6/23/2022

## **Description and Purpose of the Project**

Heavy episodic alcohol use within the college student population is widespread, creating problems for student drinkers, their peers, and their institutions. Negative consequences from heavy alcohol use can be mild (e.g., hangovers, missed classes), to severe (e.g., assault, even death). Although online interventions targeting college student drinking reduce alcohol consumption and associated problems, they are not as effective as in-person interventions. Online interventions are cost-effective, offer privacy, reduce stigma, and may reach individuals who would otherwise not receive treatment. In a recently completed randomized, controlled trial, an emailed booster with personalized feedback improved the efficacy of a popular online intervention (Braitman & Henson, 2016). Although promising, the booster incorporated in the study needs further empirical refinement.

The current project seeks to build on past progress by further developing and refining the booster. In particular, the personalized normative feedback incorporated in the booster has a strong history of empirical support, but feedback regarding protective behavioral strategies one can use to protect themselves from harm remains relatively unexplored. The current study aims to assess the added value of feedback regarding protective behavioral strategies (PBS) to emailed boosters containing personalized normative feedback (PNF). Outcomes will be compared for participants who receive a follow-up booster with PBS+PNF versus PNF alone.

There are 3 conditions: all participants receive the initial online intervention targeting college drinking. Condition 1 (the control group) receives an email with a reminder to complete the follow-up surveys, but no feedback (i.e., no booster). Condition 2 receives an emailed booster with PNF only. Condition 3 receives an emailed booster with PNF plus PBS feedback. The booster PNF content alone may be sufficiently efficacious, or the additional PBS feedback may enhance the effect.

#### **Primary Aims**

The aim of the current study is to examine if PBS feedback enhances the tailored feedback received via booster email.

#### **Participants**

Eligible participants must be 1) a current college student at the sponsor institution at the time of enrollment; 2) between the ages of 18 and 24; and 3) consumed at least one standard drink of alcohol in the past 2 weeks.

#### **Recruitment Procedure**

Recruitment uses two methods. 1) Potential participants enrolled in the sponsoring institution's psychology research pool view a brief study description. If they choose to participate, they sign up online for a timeslot to participate in the baseline session. 2) An advertisement is placed in the Announcement system at the host institution, which includes a link to a screener survey. In addition to the assessing eligibility criteria (age, student status, and alcohol consumed) additional irrelevant questions are included in the screener survey to discourage ineligible participants from re-taking the screener survey with different answers. Students who screen as eligible are invited to provide their contact information (name, email, and phone number), and to schedule their participation in the baseline session via Calendly).

### **Study Procedure**

Emerging adult college drinkers are recruited as described above. After completing the screener to verify eligibility, participants schedule their baseline session. After completing baseline, they are invited to complete two follow-up surveys 1 and 3 months after their baseline session. Participants receive a \$20 gift card (from Amazon or Target; announcements recruitment only) for baseline participation, OR their choice of a \$20 payment or credit in their course (through SONA) for baseline participation (SONA recruitment only). Additionally, participants receive \$10 for each completed follow-up survey (for the 1-, 3-month assessments). As an additional incentive, participants who complete all assessments are given a \$10 bonus (yielding \$50 total for the study if monetary compensation was chosen for the baseline protocol, and both follow-up surveys were completed).

Baseline: Upon arrival at the research lab, participants are provided with the informed consent document, and have the opportunity to ask questions. After consenting to participate, they are directed to one of the computers in the lab. Because data are collected in a computer lab setting, each computer has a privacy partition (behind and beside the monitor). This is to minimize the possibility of participants viewing each other's screens. Additionally, participants are provided with headphones to minimize disruption from the other computers. All participants complete a computerized survey at the beginning of their first appointment that assesses alcohol use, alcohol-related problems, protective behavioral strategies for drinking and their perceived effectiveness, motives and expectancies for alcohol use, anonymized social network characteristics, context of their most recent drinking occasion, marijuana and tobacco use, and demographics measures. Upon beginning the survey, participants are randomly assigned within the survey system to one of the three study conditions: neutral email (no feedback), PNF-only booster email, or PNF+PBS feedback booster email. After completing the initial assessment, participants are then directed to navigate through the eCHECKUP TO GO for Alcohol program (San Diego State University Research Foundation, 2018) until it is completed (approximately 20-30 minutes).

<u>Follow up assessments</u>: Approximately one and three months after the initial assessment, researchers send each participant an email reminding them to complete the follow-up assessment in exchange for payment. This email includes a link to an online follow-up survey that assesses alcohol use, related problems, protective behavioral strategies for drinking and their perceived effectiveness, anonymized social network characteristics, context of their most recent drinking occasion, and marijuana and tobacco use.

<u>Boosters</u>: Approximately two weeks after the intervention, all participants receive an additional email from the researcher. Information in the emails for the experimental booster groups serve as a booster to the original intervention. Baseline data are used to provide students with normative information (e.g., typical drinking among ODU students who are male/female depending on the gender of the recipient). In the PNF+PBS feedback booster group, the email also contains reminders of protective behavioral strategies they can use to reduce drinking-related harm (separated by those they reported using, versus those they have not). Participants in the control condition receive an email with no feedback.

### **Measures**

The same measures are included in baseline and the follow-up surveys:

Participants' alcohol use is assessed using a modified version of the Daily Drinking Questionnaire for the past 30 days (Collins et al., 1985). Additionally, participants describe specific aspects regarding their drinking in the past 30 days (e.g., highest consumption in a single day). Descriptive Norms are assessed by modifying the DDQ to reflect their expectations for typical male students at the same institution, typical female students at the same institution, and close friends. Injunctive Norms are assessed using 10 items (Carey et al., 2010). Alcohol-related **problems** are assessed using the 48-item Young Adult Alcohol Consequences Questionnaire (YAACQ; Read et al., 2006), modified to assess the past 30 days rather than the past year. **Protective behavioral strategy** (PBS) use is assessed using Sugarman and Carey's (2007) Strategy Questionnaire (SQ). Perceived effectiveness of PBS is assessed by modifying the instructions and response scale for Sugarman and Carey's (2007) measure to assess how effective participants perceive each strategy to be. Importance of PBS use for all people and self are assessed with 10 items created by the researcher. Alcohol expectancies are assessed using the Comprehensive Effects of Alcohol questionnaire (CEOA; Fromme et al., 1993). Motives for alcohol use are assessed using the Drinking Motives Questionnaire (DMQ; Cooper, 1994). **Alcohol beliefs** about how salient alcohol use is to college life are assessed using the College Life Alcohol Salience Scale (CLASS; Osberg et al., 2010). Social network and affiliated characteristics are assessed using the adapted version (DeMartini et al., 2013) of the Brief Important People Interview (BIPI; Zywiak et al., 2002). Participants are asked to report characteristics and context for their most recent drinking occasion. This assessment is a collection of items mostly created by the researcher, but incorporates a modified version of the Alcohol Offers scale (Read et al., 2005), and a truncated, occasion-specific version of drinking motives (Cooper, 1994). Marijuana use is assessed similar to prior research (e.g., Collins et al., 2014), and tobacco use is assessed using items created by the researcher. Demographics and general information are collected during the initial assessment only; participants report their age, race, sex, Greek affiliation (i.e., membership in fraternities or sororities), GPA, class standing, athletic status student status (full- versus part-time), residential status, relationship status, sexual identity, height, and weight (for blood alcohol content calculations).

#### References

- Braitman, A. L., & Henson, J. M. (2016). Personalized boosters for a computerized intervention targeting college drinking: The influence of protective behavioral strategies. *Journal of American College Health*, 64(7), 509-519. https://doi.org/10.1080/07448481.2016.1185725
- Carey, K. B., Henson, J. M., Carey, M. P., & Maisto, S. A. (2010). Perceived norms mediate effects of a brief motivational intervention for sanctioned college drinkers. *Clinical Psychology: Science and Practice*, *17*, 58-71. <a href="https://doi.org/10.1111/j.1468-2850.2009.01194.x">https://doi.org/10.1111/j.1468-2850.2009.01194.x</a>
- Collins, R. L., Parks, G. A., & Marlatt, G. A. (1985). Social determinants of alcohol consumption: The effects of social interaction and model status on the self-administration of alcohol. *Journal of Consulting and Clinical Psychology*, *53*(2), 189-200. https://doi.org/10.1037/0022-006X.53.2.189
- Collins, R. L., Vincent, P. C., Yu, J., Liu, L., & Epstein, L. H. (2014). A behavioral economic approach to assessing demand for marijuana. *Experimental and Clinical Psychopharmacology*, 22(3), 211-221. <a href="https://doi.org/10.1037/a0035318">https://doi.org/10.1037/a0035318</a>
- Cooper, M. L. (1994). Motivations for alcohol use among adolescents: Development and validation of a four-factor model. *Psychological Assessment*, *6*(2), 117–128. https://doi.org/10.1037/1040-3590.6.2.117
- Core Institute. (2006). American Campuses: 2006 Statistics on Alcohol and Other Drug Use. Carbondale, IL: Southern Illinois University.
- DeMartini, K. S., Prince, M. A., & Carey, K. B. (2013). Identification of trajectories of social network composition change and the relationship to alcohol consumption and norms. *Drug and Alcohol Dependence*, *132*, 309-315.

  <a href="https://doi.org/10.1016/j.drugalcdep.2013.02.020">https://doi.org/10.1016/j.drugalcdep.2013.02.020</a>
- Fromme, K., Stroot, E. A., & Kaplan, D. (1993). Comprehensive effects of alcohol: Development and psychometric assessment of a new expectancy questionnaire. *Psychological Assessment*, *5*(1), 19-26. https://doi.org/10.1037/1040-3590.5.1.19
- Muthén, L. K., & & Muthén, B. O. (1998-2017). *Mplus User's Guide* (8 edition). Muthén & Muthén.
- Osberg, T. M., Atkins, L., Buchholz, L., Shirshova, V., Swiantek, A., Whitley, J., et al. (2010). Development and validation of the College Life Alcohol Salience Scale: A measure of beliefs about the role of alcohol in college life. *Psychology of Addictive Behaviors*, 24(1),1–12. <a href="https://doi.org/10.1037/a0018197">https://doi.org/10.1037/a0018197</a>
- Read, J. P., Kahler, C. W., Strong, D. R., & Colder, C. R. (2006). Development and preliminary validation of the Young Adult Alcohol Consequences Questionnaire. *Journal of Studies on Alcohol*, 67(1), 169-177. https://doi.org/10.15288/jsa.2006.67.169
- Read, J. P., Wood, M. D., & Capone, C. (2005). A prospective investigation of relations between social influences and alcohol involvement during the transition into college. *Journal of Studies on Alcohol*, 66, 23–34. <a href="https://doi.org/10.15288/jsa.2005.66.23">https://doi.org/10.15288/jsa.2005.66.23</a>
- San Diego State University Research Foundation. (2018). eCHECKUP TO GO [Online program]. http://www.echeckuptogo.com/programs/alcohol
- Scott-Sheldon, L. A. J., Carey, K. B., Elliott, J. C., & Garey, L., & Carey, M P. (2014). Efficacy of alcohol interventions for first-year college students: A meta-analytic review of randomized controlled trials. *Journal of Consulting and Clinical Psychology*, 82(2), 177-188. https://doi.org/10.1037/a0035192

- Sugarman, D. E., & Carey, K. B. (2007). The relationship between drinking control strategies and college student alcohol use. *Psychology of Addictive Behaviors*, 21(3), 338-345. <a href="https://doi.org/10.1037/0893-164x.21.3.338">https://doi.org/10.1037/0893-164x.21.3.338</a>
- Zwyiak, W. H., & Longabaugh, R. (2002). *The Brief Important People Interview Manual*. Center for Alcohol and Addiction Studies, Providence, RI.